CLINICAL TRIAL: NCT07239817
Title: PENG 360°: PENG Block + LIA Nella Endoprotesi di Anca Con Accesso Anteriore.
Brief Title: PENG Block + LIA For Endoprosthesis Surgery With Anterior Approach
Acronym: PENG 360°
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Romualdo Del Buono, Principal Investigator, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PeBILIA 5680-25.06.2025
Record Dates: First submitted 2025-09-30; First posted 2025-11-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures; Arthroplasty, Replacement, Hip; Pain, Postoperative; Anesthesia and Analgesia; Nerve Block; Local Anesthesia Infiltration
Keywords: Pericapsular Nerve Group Block; PENG block; Local Infiltration Analgesia; Spinal Anesthesia; Hip Arthroplasty; Postoperative Pain; Femoral Fractures; Ultrasound Guidance; Early Mobilization
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative; Agnosia; Femoral Fractures | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG 360° (Experimental): Participants assigned to this arm will receive a motor-sparing anesthetic technique. This consists of three ultrasound-guided injections performed before surgery: an anterior Pericapsular Nerve Group (PENG) block, a Local Infiltration Analgesia (LIA) of the incision line, and a posterior PENG (PONG) block.
  Interventions: Procedure: Pericapsular Nerve Group Blocks with Local Infiltration Analgesia
- Spinal (Active Comparator): Participants assigned to this arm will receive standard spinal anesthesia. The procedure will be performed according to the center's standard practice and guidelines, with the choice of local anesthetic and dosage at the discretion of the anesthesiologist
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Blocks with Local Infiltration Analgesia — An ultrasound-guided, motor-sparing regional anesthesia procedure. It involves three distinct injections: 1) An anterior Pericapsular Nerve Group (A-PENG) block targeting the sensory articular branches of the femoral and obturator nerves. 2) A Local Infiltration Analgesia (LIA) of the surgical incision line. 3) A posterior PENG (PONG) block targeting sensory branches from the sciatic plexus. The local anesthetic mixture consists of ropivacaine, mepivacaine with epinephrine, and dexamethasone in specific volumes for each injection site.
  Other Names: PENG 360°; A-PENG +PONG +LIA
  Arms: PENG 360°
Procedure: spinal anesthesia — Standard neuraxial anesthesia technique involving the injection of a local anesthetic into the subarachnoid space. The procedure is performed according to the institution's standard clinical practice. The choice of the specific local anesthetic agent, dose, and technique will be at the discretion of the attending anesthesiologist, based on the participant's clinical characteristics.
  Other Names: Spinal Block; Subarachnoid Block
  Arms: Spinal

SUMMARY:
The goal of this clinical trial is to learn if a new local anesthesia technique can control pain as well as the standard spinal anesthesia for adults having hip endoprosthesis surgery. The main questions it aims to answer are:

* Is the new local anesthesia technique as effective as standard spinal anesthesia in managing pain during the first two days after surgery?
* Does the new technique allow participants to move their leg sooner after the operation?

Researchers will compare the new local anesthesia technique (numbing medicine injected directly around the hip joint) to standard spinal anesthesia (a numbing injection in the back) to see if the new technique works just as well for pain control while possibly causing fewer side effects like nausea.

Participants who join this study will be randomly placed into one of two groups.

One group will receive the standard spinal anesthesia before their surgery.

The other group will receive the new local anesthesia technique before their surgery.

After the operation, researchers will track the amount of extra pain medicine each participant uses and will check their ability to move their hip, knee, and foot.

DETAILED DESCRIPTION:
Study Rationale Standard anesthetic techniques for hip fracture surgery in the target population, which often includes fragile and elderly individuals, present distinct challenges. Both neuraxial (spinal) and general anesthesia can have a significant hemodynamic impact. Furthermore, traditional regional anesthetic techniques like lumbar plexus or femoral nerve blocks, while providing effective analgesia, often result in significant motor and sensory blockade of the lower limb, which can impede early mobilization and rehabilitation.

This study investigates a motor-sparing anesthetic approach. The intervention is based on pericapsular nerve group blocks (A-PENG and PONG), anterior and posterior, which target only the sensory articular branches innervating the hip capsule. This technique, combined with local infiltration analgesia (LIA), aims to provide comprehensive surgical anesthesia and post-operative analgesia without affecting motor function, thereby facilitating immediate post-operative mobilization.

Anesthetic Intervention Details (PENG 360° Arm) Participants randomized to the investigational arm will receive a combination of three injections prior to surgical incision. A convex ultrasound probe will be used for A-PENG and PONG.

* Anterior A-PENG Block: An injection of 20 mL of "plain" anesthetic solution is administered into the fascial plane between the iliopsoas muscle and the hip joint capsule. This solution consists of 10 mL of 0.75% ropivacaine, 10 mL of 2% mepivacaine with 1:200,000 epinephrine, and 2 mg of dexamethasone.
* Local Infiltration Analgesia (LIA): An injection of 20 mL of "diluted" anesthetic solution is used to infiltrate the planned incision line and subcutaneous tissue. This solution consists of 5 mL of 0.75% ropivacaine, 5 mL of 2% mepivacaine with 1:200,000 epinephrine, 1 mg of dexamethasone, and 10 mL of normal saline.
* Posterior PONG Block: With the participant in the lateral decubitus position, an injection of 10 mL of "plain" anesthetic solution is administered into the fascial plane deep to the quadratus femoris muscle. This solution consists of 5 mL of 0.75% ropivacaine, 5 mL of 2% mepivacaine with 1:200,000 epinephrine, and 1 mg of dexamethasone.

During surgery, participants in this arm will receive supplemental oxygen and sedation with propofol, with the depth of anesthesia monitored using a Bispectral Index (BIS) monitor.

Post-operative Pain Management Protocol To ensure a standardized approach to analgesia for all participants in both study arms, a uniform post-operative pain management protocol will be implemented. Unless contraindicated, all participants will receive a fixed-dose regimen of intravenous paracetamol (1000 mg) and ketorolac (30 mg) every 8 hours.

In addition, all participants will be provided with an intravenous patient-controlled analgesia (PCA) pump delivering morphine. The PCA pump will be set to deliver on-demand rescue boluses of 2 mg of morphine with no continuous background infusion. The maximum daily dose will be limited to 10 mg for participants over 65 years of age and 20 mg for those 65 or younger.

Data Management and Randomization Participant data will be collected and managed using an electronic Case Report Form (CRF) built with Google Forms and stored in a secure cloud database (Google Sheets). All data will be pseudonymized using a unique alphanumeric identifier assigned at the time of enrollment to ensure participant confidentiality.

Randomization will be performed using a dedicated Google Form configured to provide response options in a random order. The investigator will select the first option presented to assign the participant to either the "case" or "control" group19.

Statistical Analysis Plan Descriptive statistics (mean, median, standard deviation, min/max) will be used to summarize the collected data. The primary endpoint (cumulative number of PCA rescue doses at 48 hours) will be analyzed using a Poisson distribution model.

For other outcomes, a Chi-square test will be used for categorical variables (e.g., need for conversion to general anesthesia), while a t-test (or a non-parametric equivalent) will be used for continuous variables (e.g., NRS pain scores in the recovery room). Analysis of covariance and multiple linear regression may also be conducted to evaluate the role of demographic and clinical characteristics on study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Scheduled for hip endoprosthesis surgery for femoral fracture with an anterior approach.
* Age 18 years or older.
* Willing and able to comply with the study protocol.

Exclusion Criteria:

* Failure to provide informed consent.
* Age less than 18 years.
* Known allergy to local anesthetics or other medications used in the protocol.
* Presence of infection at the planned injection site.
* Pre-existing hip prosthesis or prior major surgery on the same hip (e.g., revision surgery).
* ASA physical status class > IV.
* Administration of intraoperative opiates or conversion to general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Postoperative Analgesic Rescue Doses | From arrival in the Post-Anesthesia Care Unit (PACU) up to 48 hours after surgery.
  The cumulative number of on-demand analgesic doses (2 mg morphine bolus) requested by the participant via an intravenous Patient-Controlled Analgesia (PCA) pump. The total number of requests will be recorded from the pump's memory at 48 hours postoperatively. This is the primary measure for assessing postoperative pain control.

SECONDARY OUTCOMES:
Immediate Postoperative Limb Mobility | Upon arrival in the Post-Anesthesia Care Unit (PACU), approximately 0-1 hours after surgery.
  Assessment of motor function in the operated limb. A binary (Yes/No) assessment will be made of the participant's ability to actively move their hip, knee, and foot.
Incidence of Postoperative Nausea and Vomiting (PONV) | Within the first 48 hours after surgery.
  The occurrence of any episode of nausea or vomiting as reported by the participant or observed by clinical staff will be recorded.
Postoperative Pain Intensity | Upon arrival in the Post-Anesthesia Care Unit (PACU), approximately 0-1 hours after surgery.
  Participant's self-reported pain intensity will be measured using the Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable.
Length of Hospital Stay | From the date of surgery until date of hospital discharge, assessed up to 30 days.
  The total number of days from the day of surgery to the day of discharge from the hospital, which is an indirect measure of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Romualdo Del Buono, MD, Principal Investigator — Unit of Anesthesia, Intensive Care and Pain Management, ASST Gaetano Pini, Milan, Italy;
Locations (1):
- Gaetano Pini-CTO, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Plan Description
  Individual Participant Data (IPD) that will be shared:
  The full, de-identified participant dataset.
  The final study protocol.
  The statistical analysis plan.
  How to access the data:
  Data will be available to qualified researchers for non-commercial, academic purposes upon reasonable request. Interested researchers should submit a formal proposal outlining their research goals to the Principal Investigator.
  Data sharing timeline:
  Data will be made available after the publication of the primary study results and will remain available for a period of 5 years.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available starting 6 months after the publication of the primary manuscript. Data will remain available for a period of 5 years following publication.
Access Criteria: Access to the de-identified individual participant data and supporting documents will be granted to qualified academic researchers for non-commercial purposes, such as secondary analysis or meta-analysis. Researchers must submit a formal research proposal to the Principal Investigator for review. A signed data sharing agreement will be required before data is transferred.

REFERENCES:
- [Background] Del Buono R, Pascarella G, Costa F, Barbara E. Ultrasound-guided local infiltration analgesia for hip surgery: myth or reality? Minerva Anestesiol. 2019 Nov;85(11):1242-1243. doi: 10.23736/S0375-9393.19.13701-7. Epub 2019 May 21. No abstract available. PMID 31124626
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular nerve group block: an overview. Minerva Anestesiol. 2021 Apr;87(4):458-466. doi: 10.23736/S0375-9393.20.14798-9. Epub 2021 Jan 12. PMID 33432791
- [Background] Del Buono R, Pascarella G, Padua E, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. PENG block: from standard to unconventional approaches. Minerva Anestesiol. 2021 Oct;87(10):1157-1158. doi: 10.23736/S0375-9393.21.15847-X. Epub 2021 Jul 14. No abstract available. PMID 34263587
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Reply to: Tips for pericapsular nerve group (PENG) neurolytic blocks. Minerva Anestesiol. 2021 Oct;87(10):1151-1152. doi: 10.23736/S0375-9393.21.16019-5. Epub 2021 Aug 2. No abstract available. PMID 34337929
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular hip radiofrequency: future approaches to treat hip chronic pain. Minerva Anestesiol. 2021 Dec;87(12):1393-1394. doi: 10.23736/S0375-9393.21.16081-X. Epub 2021 Sep 16. No abstract available. PMID 34527412
- [Background] Del Buono R, Tognu A. Hip replacement using pericapsular nerve blocks in a high-risk patient. Minerva Anestesiol. 2024 Nov;90(11):1052-1054. doi: 10.23736/S0375-9393.24.18242-9. Epub 2024 Jul 9. No abstract available. PMID 38980297
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657